CLINICAL TRIAL: NCT04059003
Title: Circulating Tumor Cell Changes and Efficacy of Neoadjuvant Chemotherapy for Triple-negative Breast Cancer: a Cohort Trial
Brief Title: CTC Changes and Efficacy of Neoadjuvant Chemotherapy for Triple-negative Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Jianyi Li, Principal Investigator, Shengjing Hospital
Other Study IDs: Shengjing-LJY03
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Breast Neoplasms
Keywords: Biomarkers; Tumor; Positron Emission Tomography; Computed Tomography
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sensitivity group: 100 patients will be assigned into sensitivity group according to the actual situation of them.
  Interventions: Drug: Taxanes or/and anthracycline-based therapy
- Drug resistance group: 100 patients will be assigned into drug resistance according to the actual situation of them.
  Interventions: Drug: Taxanes or/and anthracycline-based therapy

INTERVENTIONS:
Drug: Taxanes or/and anthracycline-based therapy — Taxanes or/and anthracycline-based therapy will be used in this group. That is, intravenous injection of 90 mg/m2 epirubicin (trade name: Pharmorubicin, Pfizer, Shanghai, China; drug approval number: H20100155) + 135 mg/m2 paclitaxel liposome (trade name: Taxotere, Sanofi (Hangzhou) Pharmaceutical Co., Ltd., Hangzhou, China; drug approval number: J20090104), every 3 weeks as a course of treatment. The efficacy will be evaluated every 2 courses. After the 6th course, mastectomy will be performed according to the patient's conditions.

SUMMARY:
Chemotherapy before operation for malignant tumors can reduce the size of tumors to a certain extent, even eliminate micrometastases. Chemotherapy can also detect the sensitivity of chemotherapeutic drugs and create opportunities for breast-conserving or surgical treatment for patients. This may lead to high survival opportunities for triple-negative breast cancer patients who are not sensitive to targeted therapy or endocrine therapy. However, during neoadjuvant therapy, CT or MRI tests are needed to monitor the patient's condition. Therefore, if there is any deterioration, to consider changing the treatment regimen or immediately carrying out surgery is necessary. However, because of the need for multiple imaging examinations during neoadjuvant therapy, which will increase medical costs, to explore a cheaper examination method is necessary . Circulating tumor cells in peripheral blood are derived from the shedding of breast cancer lesions. Detection of these circulating tumor cells may monitor the therapeutic effect on breast cancer, and the cost of detecting circulating tumor cells is much lower than that of conventional PET-CT, which can obviously reduce the medical costs of patients. However, there is no clinical study on the changes of circulating tumor cells and the efficacy of neoadjuvant chemotherapy in the treatment of triple-negative breast cancer in and outside China.

DETAILED DESCRIPTION:
Triple-negative breast cancer refers to breast cancer with negative human epidermal growth factor receptor 2, estrogen receptor and progesterone receptor. Triple-negative breast cancer has poor differentiation, high invasiveness and high recurrence rate, accounting for 15.0%-23.8% of breast cancer. Due to the phenotypic specificity of triple-negative breast cancer, both targeted therapy and endocrine therapy are insensitive, making chemotherapy an important part in the treatment of triple-negative breast cancer.

In 1982, Frei proposed the concept of neoadjuvant chemotherapy, which is to apply chemotherapy before surgery for malignant tumors. Chemotherapy can reduce the size of tumors to some extent, even eliminate micrometastases, detect the sensitivity of chemotherapy drugs, and create opportunities for patients to have breast-conserving or surgical treatment. For triple-negative breast cancer, neoadjuvant chemotherapy with synchronous combination of anthracyclines and taxanes or intensive sequential combination of anthracyclines and taxanes is the first choice. Simultaneously, chemotherapeutic drugs such as platinum, albumin, and paclitaxel as well as poly-ADP-ribose polymerase inhibitors can be added according to the patient's condition. However, during neoadjuvant therapy, a CT or MRI test is needed to monitor the patient's condition, so if there is any deterioration, to consider changing the treatment plan or immediately performing surgery is necessary. However, because of the need for multiple imaging examinations during neoadjuvant therapy, which increases the medical costs, to explore a low cost inspection method is necessary.

Circulating tumor cells are a new type of tumor molecular marker. Circulating tumor cells in peripheral blood originate from breast cancer (primary and metastatic lesions) shedding. Detection of these circulating tumor cells may monitor the therapeutic effect on breast cancer. The cost of detecting circulating tumor cells is much lower than that of conventional PET-CT, which can noticeably reduce medical expenses of patients. However, there is no clinical study on the changes of circulating tumor cells and the efficacy of neoadjuvant chemotherapy for triple-negative breast cancer in and outside China. This study aims to explore the correlation between the changes of circulating tumor cells and the efficacy of neoadjuvant chemotherapy for triple-negative breast cancer, and to compare the time intervals between the changes of circulating tumor cells and the changes of efficacy in patients with different sensitivities of neoadjuvant chemotherapy, so as to provide experimental evidence for predicting the efficacy of neoadjuvant chemotherapy by observing the changes of circulating tumor cells in clinic.

ELIGIBILITY:
Inclusion Criteria:

* triple-negative breast cancer confirmed by breast biopsy;
* stage III breast cancer (IIIA-C) assessed by CT or MRI;
* neoadjuvant chemotherapy;
* informed consent of patients and their family members.

Exclusion Criteria:

* use of second-line chemotherapy regimen;
* bilateral breast cancer;
* inflammatory breast cancer;
* pregnant or breast-feeding;
* distant metastasis;
* a history of other cancers or chest radiotherapy;
* a history of abnormal blood test or other infectious symptoms.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Totally 200 patients who meet the inclusion and exclusion criteria will be consecutively enrolled in the trial and grouped according to their sensitivity.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of neoadjuvant chemotherapy | At 18 weeks
  The efficacy will be evaluated by the response evaluation criteria in solid tumors (RECIST) score, which is based on CT or X-ray results. (1) Complete response (CR): disappearance of all lesions; (2) partial response (PR): 30% decrease in sum of all target lesions in longest axis measurement; (3) stable disease (SD): the sum of the longest diameter of all lesions decreases but does not reach PR or increases but does not reach PD; (4) progressive disease (PD): 20% increase in the sum of the longest diameter or appearance of new lesions. SD: One or more non-target lesions and/or tumor markers are higher than normal and persistent.

SECONDARY OUTCOMES:
Efficacy of neoadjuvant chemotherapy | At 6 and 12 weeks
  The efficacy will be evaluated by the response evaluation criteria in solid tumors (RECIST) score, which is based on CT or X-ray results. (1) Complete response (CR): disappearance of all lesions; (2) partial response (PR): 30% decrease in sum of all target lesions in longest axis measurement; (3) stable disease (SD): the sum of the longest diameter of all lesions decreases but does not reach PR or increases but does not reach PD; (4) progressive disease (PD): 20% increase in the sum of the longest diameter or appearance of new lesions. SD: One or more non-target lesions and/or tumor markers are higher than normal and persistent.
Detection of circulating tumor cells | At 3 weeks of neoadjuvant chemotherapy
  At 3 weeks of neoadjuvant chemotherapy, 2.5 ml of blood will be taken from median elbow vein of upper arm, and the number of circulating tumor cells is ≤ 2 or CD133 ≤ 1.
Miller-Payne grading score | Before and 18 weeks after chemotherapy
  The Miller-Payne grading system is as follows: Grade 1: no reduction in overall cellularity; grade 2: up to 30% reduction of cellularity; grade 3: between an estimated 30% and 90% reduction in tumor cellularity; grade 4: a marked disappearance of more than 90% of tumor cells; grade 5: no invasive malignant cells identifiable in sections from the site of the tumor, but ductal carcinoma in situ may be present.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyi Li, Principal Investigator — Shengjing Hospital
Locations (2):
- China (2):
  - Cancer Hospital of China Medical University, Liaoning Cancer Hospital and Institute, Shengyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning